CLINICAL TRIAL: NCT02577679
Title: Associations Between Periodontitis and Autoimmune Antibodies in Rheumatoid Arthritis Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201503116RINA
Record Dates: First submitted 2015-09-23; First posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Periodontitis, Rheumatoid Arthritis, Autoimmunity,
Keywords: Dentistry
MeSH Terms: conditions — Periodontitis; Arthritis, Rheumatoid; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this case control study is to explore the possible association between periodontal destruction and serum anti-CCP antibodies in RA patients and healthy subjects.

DETAILED DESCRIPTION:
In patients with RA, the anti-CCP antibody titer seems positively correlated to their periodontal destruction and disease activity in comparison with healthy subjects.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physically healthy persons, especially free of any autoimmune diseases, DM, CVD. No history of periodontal treatment.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Serum level of anti-cyclic citrullinated peptide/protein antibody | Base line
  Lower then 7 Unit/milliliter: negative 7-10 Unit/milliliter: weak positive Higher then 10 Unit/milliliter: positive
Periodontal pocket depth and clinical attachment level | Baseline
  Lower then 4 millimeter: normal Higher then 4 millimeter: diseased/previously diseased

SECONDARY OUTCOMES:
Serum level of tumor necrotic factor alpha | Baseline
  Recorded in picogram per milliliter
Serum level of anti-mutated citrullinated vimentin | Baseline
  Recorded in Unit per milliliter
Serum level of interleukin 6 | Baseline
  Recorded in picogram per milliliter
Serum level of interleukin 17 | Baseline
  Recorded in picogram per milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Wen Chen, PhD, Study Director — Assistant professor
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan